CLINICAL TRIAL: NCT01867606
Title: MC1267, A Randomized, Blinded Pilot Placebo-Controlled Trial With Oral Serum Bovine Immunoglobulin (SBI) to Assess Quality of Life and the Faster Post-Operative Recovery of Gynecological Cancer Patients
Brief Title: Serum Bovine Immunoglobulin Protein Isolate in Improving Quality of Life and Post-Operative Recovery in Patients With Gynecological Cancer After Undergoing Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MC1267; NCI-2013-00866 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1267 (Other: Mayo Clinic); 12-009448 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2013-05-29; First posted 2013-06-04 (Estimated); Results first posted 2020-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Female Reproductive Cancer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (serum-derived bovine immunoglobulin protein isolate) (Experimental): Patients receive SBI PO BID on days 1-28.
  Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: serum-derived bovine immunoglobulin protein isolate; Other: laboratory biomarker analysis; Other: quality-of-life assessment; Other: questionnaire administration
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO BID on days 1-28.
  Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: placebo; Other: laboratory biomarker analysis; Other: quality-of-life assessment; Other: questionnaire administration

INTERVENTIONS:
Biological: serum-derived bovine immunoglobulin protein isolate — Given PO
  Other Names: SBI; serum bovine immunoglobulin
  Arms: Arm I (serum-derived bovine immunoglobulin protein isolate)
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: laboratory biomarker analysis — Correlative studies
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary studies

SUMMARY:
This randomized pilot phase II trial studies how well serum bovine immunoglobulin protein isolate works in improving quality of life and post-operative recovery in patients with cancer of the female reproductive tract after undergoing surgery. Serum bovine immunoglobulin may help provide nutrition to patients who are not able to eat or digest ordinary food. This may improve the quality of life of patients with gynecological cancer and help them recover more quickly from surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the time-to-quality of life (QOL) improvement from baseline in postoperative gynecological cancer patients who are receiving oral serum bovine immunoglobulin (SBI) vs. placebo.

SECONDARY OBJECTIVES:

I. To compare the surgical complication rates between oral SBI vs. placebo up to 1 month post-surgery (safety endpoint).

II. To compare the QOL, as derived from the previously-validated Symptom Distress Scale, the Postoperative Quality of Life questionnaire (PQL), and the uniscale (overall QOL item) between patients receiving oral SBI vs. placebo.

III. To compare the grade 2 or worse adverse event rates for patients receiving oral SBI vs. placebo.

IV. To characterize the adverse event profile of oral SBI in postoperative gynecological cancer patients (safety endpoint).

V. To compare supplement adherence between patients receiving oral SBI vs. placebo.

TERTIARY OBJECTIVES:

I. To explore whether candidate biomarkers are modified with SBI versus placebo.

II. As part of ongoing research, to bank leftover blood samples for future studies.

III. To explore quality of life during postoperative recovery after gynecologic surgery, regardless of whether or not patients take the study intervention/placebo or discontinue intervention/placebo early.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive SBI orally (PO) twice daily (BID) on days 1-28.

ARM II: Patients receive placebo PO BID on days 1-28.

In both arms, treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gynecological cancer of any type or strong suspicion for cancer
* Patients must have begun postoperative oral intake of food prior to registration
* Open laparotomy or laparoscopic surgery undertaken with cancer therapeutic intent (not a subsequent surgery to manage a postoperative complication) that had occurred =< 7 days prior to registration and that entailed more than a simple hysterectomy
* Creatinine =< 1.5 x the upper limit of normal (ULN)
* Absolute neutrophil count >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide informed written consent
* Negative (serum) pregnancy test done =< 7 days prior to randomization, for women of childbearing potential only
* Willing to provide mandatory baseline blood samples for correlative research purposes

Exclusion Criteria:

* Symptomatic and/or untreated brain metastases
* Ongoing parenteral nutrition (receiving intravenous nutrition support at the time of enrollment); note: patients may be receiving maintenance intravenous (IV) fluids
* Current enrollment in any other trial that entails the concurrent administration of any other agent designed to enhance postoperative recovery
* Allergy to beef

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-10-04 (Actual); Primary Completion 2015-11-21 (Actual); Study Completion 2015-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Serum-derived Bovine Immunoglobulin Protein Isolate): Patients receive SBI PO BID on days 1-28.>>
  >> Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.>>
  >> serum-derived bovine immunoglobulin protein isolate: Given PO>>
  >> laboratory biomarker analysis: Correlative studies>>
  >> quality-of-life assessment: Ancillary studies>>
  >> questionnaire administration: Ancillary studies
- Arm II (Placebo): Patients receive placebo PO BID on days 1-28.>>
  >> Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.>>
  >> placebo: Given PO>>
  >> laboratory biomarker analysis: Correlative studies>>
  >> quality-of-life assessment: Ancillary studies>>
  >> questionnaire administration: Ancillary studies
Period: Overall Study
Arm/Group | Arm I (Serum-derived Bovine Immunoglobulin Protein Isolate) | Arm II (Placebo)
Started | 26 | 32
Completed | 16 | 17
Not Completed | 10 | 15
Not completed — Withdrawal by Subject | 10 | 14
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm II (Placebo) | Arm I (Serum-derived Bovine Immunoglobulin Protein Isolate) | Total
Number analyzed (Participants) | 32 | 26 | 58
Age, Continuous [Median (Full Range); unit: Years] | 62 [32 to 81] | 62 [37 to 79] | 62 [32 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 26 | 58
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 29 | 24 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Time-to-QOL Improvement Defined as Any Increase in the QOL Score Measured Using the Total Score of the 14-item Postoperative Quality of Life (PQL) Tool
Description: For this endpoint, the total QOL score could range from 1 to 140 (0 being the worst and 140 being the best). The primary analysis will be a comparison of oral SBI vs. placebo using a two-sided log-rank test between the 2 Kaplan-Meier curves.the total score of the 14-item Postoperative Quality of Life (PQL) tool [15] will be used, where the total score could range from 0 to 140 (0 being the worst and 140 being the best). These scores will be converted to the percentage scale, where a score of 140 will be converted to 100 and a score of 0 will remain as 0. This QOL will be measured weekly for the entire 12 week length of the study and at the end of the intervention. QOL improvement will be defined as at least a 10 point increase in the QOL score from baseline, on the percentage scale.
Time Frame: up to 25 months
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm I (Serum-derived Bovine Immunoglobulin Protein Isolate): Patients receive SBI PO BID on days 1-28. >
  >
  >
  >
  >
  > Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  >
  >
  >
  >
  >
  > serum-derived bovine immunoglobulin protein isolate: Given PO
- Arm II (Placebo): Patients receive placebo PO BID on days 1-28. >
  >
  >
  >
  >
  > Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  >
  >
  >
  >
  >
  > placebo: Given PO
Arm/Group | Arm I (Serum-derived Bovine Immunoglobulin Protein Isolate) | Arm II (Placebo)
Number analyzed (Participants) | 16 | 17
Months | 4.86 [3.0 to 6.43] | 3.29 [2.43 to 10.43]

2. Secondary Outcome: Overall Adverse Event Rates for Grade 2 or Higher Adverse Events, Graded According to the Common Terminology Criteria for Adverse Events Version 4.0
Description: Frequency tables will be reviewed to determine adverse event patterns, this data is reported in the adverse events section of this report. Below is the number of patients that experienced an adverse event greater than or equal to 2.
Time Frame: up to 25 months
Population: All evaluable patients
Measure: Count of Participants; unit: Participants
Groups:
- Arm I (Serum-derived Bovine Immunoglobulin Protein Isolate): Patients receive SBI PO BID on days 1-28. >>
  >> Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  >>
  >> serum-derived bovine immunoglobulin protein isolate: Given PO
- Arm II (Placebo): Patients receive placebo PO BID on days 1-28. >>
  >> Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  >>
  >> placebo: Given PO
Arm/Group | Arm I (Serum-derived Bovine Immunoglobulin Protein Isolate) | Arm II (Placebo)
Number analyzed (Participants) | 16 | 17
Participants | 5 | 10

3. Secondary Outcome: Surgical Complication Rates
Description: Compared between the 2 arms using Chi-Square or Fisher's Exact tests.
Time Frame: Up to 1 month post-surgery
Population: All evaluable patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Serum-derived Bovine Immunoglobulin Protein Isolate) | Arm II (Placebo)
Number analyzed (Participants) | 16 | 17
Participants
  Severe Complication | 3 | 3
  Moderate Complication | 2 | 7
  Mild Complication | 10 | 6
  No Complication | 1 | 1
Statistical Analysis 1: Comparison: Arm I (Serum-derived Bovine Immunoglobulin Protein Isolate) vs Arm II (Placebo); Test type: Superiority; p = 0.29, Fisher Exact

4. Secondary Outcome: Intervention Compliance Assessed Using the Compliance Questionnaire
Description: The frequency and percentage for each Compliance Questionnaire category will be summarized descriptively by cycle and by intervention arm. In addition, cycle by cycle compliance data will be compared between the 2 arms using a Chi-square test.
Time Frame: up to 25 months
Measure: Count of Participants; unit: Participants
Groups:
- Arm I (Serum-derived Bovine Immunoglobulin Protein Isolate): Patients receive SBI PO BID on days 1-28. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity. serum-derived bovine immunoglobulin protein isolate: Given PO
- Arm II (Placebo): Patients receive placebo PO BID on days 1-28. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.placebo: Given PO
Arm/Group | Arm I (Serum-derived Bovine Immunoglobulin Protein Isolate) | Arm II (Placebo)
Number analyzed (Participants) | 16 | 17
Participants
  Cycle 1: Always to Usually Compliant | 8 | 13
  Cycle 1: Occasionally to Never Compliant | 5 | 4
  Cycle 1: Missing | 3 | 0
  Cycle 1: Patient off treatment (NA) | 0 | 0
  Cycle 2: Always to Usually Compliant | 3 | 7
  Cycle 2: Occasionally to Never Compliant | 1 | 0
  Cycle 2: Missing | 0 | 1
  Cycle 2: Patient off treatment (NA) | 12 | 9

5. Secondary Outcome: Change in QOL Measured Using the 14-item PQL Tool, Uniscale, and the Previously-validated Symptom Distress Scale
Description: All 14 of the individual items from the PQL tool, along with the 4 additional items after the PQL questions will be analyzed and compared between the 2 intervention arms. Differences between post-randomization and baseline QOL scores will be analyzed and compared between the 2 arms using a Wilcoxon Rank-sum test. Also, other graphical and statistical methods will be used to compare the QOL between the 2 arms over time. For this endpoint, the total QOL score could range from 1 to 140 (0 being the worst and 140 being the best). These scores will be converted to the percentage scale, where a score of 140 will be converted to 100 and a score of 0 will remain as 0. This QOL will be measured weekly for the entire 12 week length of the study and at the end of the intervention. QOL improvement will be defined as at least a 10 point increase in the QOL score from baseline, on the percentage scale.
Time Frame: up to 25 months
Population: All evaluable patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Serum-derived Bovine Immunoglobulin Protein Isolate) | Arm II (Placebo)
Number analyzed (Participants) | 16 | 17
Participants
  Improvement | 11 | 13
  No Improvement | 5 | 4
Statistical Analysis 1: Comparison: Arm I (Serum-derived Bovine Immunoglobulin Protein Isolate) vs Arm II (Placebo); Test type: Superiority; p = 0.62, Chi-squared

6. Secondary Outcome: Change in QOL in Patients Who do Not Start Intervention or Discontinue Early, Measured Using the 14-item PQL Tool, Uniscale, and the Previously-validated Symptom Distress Scale
Description: Analysis will be descriptive in nature to see if these patients have a poorer QOL than patients who stay on study.
Time Frame: Baseline up to 25 months
Population: All evaluable patients who never started intervention or discontinue early. All patients completed the study, no patients are evaluable for this outcome.
Arm/Group | Arm I (Serum-derived Bovine Immunoglobulin Protein Isolate) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 25 months
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 were utilized for AE reporting. Participants who did NOT withdraw ("Withdrawal by Subject") from the study are included in this analysis.
Arm/Group | Arm II (Placebo) | Arm I (Serum-derived Bovine Immunoglobulin Protein Isolate)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 3/16 | 3/18
Other Adverse Events (participants affected / at risk) | 15/16 | 15/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm II (Placebo) (N=16) | Arm I (Serum-derived Bovine Immunoglobulin Protein Isolate) (N=18)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm II (Placebo) (N=16) | Arm I (Serum-derived Bovine Immunoglobulin Protein Isolate) (N=18)
Abdominal pain (Gastrointestinal disorders) | 9 (12) | 7 (16)
Bloating (Gastrointestinal disorders) | 8 (12) | 4 (7)
Diarrhea (Gastrointestinal disorders) | 4 (6) | 4 (6)
Flatulence (Gastrointestinal disorders) | 6 (7) | 9 (21)
Nausea (Gastrointestinal disorders) | 7 (8) | 8 (12)
Vomiting (Gastrointestinal disorders) | 4 (4) | 5 (5)
Fatigue (General disorders) | 12 (20) | 14 (31)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-05-07): https://cdn.clinicaltrials.gov/large-docs/06/NCT01867606/Prot_SAP_000.pdf
  • Informed Consent Form (2015-04-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT01867606/ICF_001.pdf